CLINICAL TRIAL: NCT02027012
Title: Treatment of Resistant Hypertension Using a Radiofrequency Percutaneous Transluminal Angioplasty Catheter in China
Brief Title: Treatment of Resistant Hypertension by Renal Denervation in China
Acronym: REDUCE-HTN-CN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: company strategic change
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S6007
Record Dates: First submitted 2014-01-01; First posted 2014-01-03 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Medication-resistant Hypertension

STUDY DESIGN:
Intervention Model Description: Vessix device
Oversight: Data Monitoring Committee: No

ARMS (1):
- Renal denervation with Vessix system (Experimental)
  Interventions: Device: Percutaneous renal denervation with the Vessix™ Renal Denervation System

INTERVENTIONS:
Device: Percutaneous renal denervation with the Vessix™ Renal Denervation System
  Other Names: Vessix Renal Denervation System

SUMMARY:
REDUCE-HTN-China study is a prospective, multi-center, single cohort study for the percutaneous therapeutic treatment of medication-resistant hypertension in China.The primary objective is to assess the efficacy performance of the Vessix™ Renal Denervation System for the treatment of medication resistant hypertension on the basis of the hypothesis that the percutaneous therapeutic renal denervation for the treatment of medication-resistant hypertension using the Vessix™ Renal Denervation System will reduce systolic (SBP) and diastolic blood pressure (DBP) at 6- month compared to baseline as accessed by office-based blood pressure measurements.

DETAILED DESCRIPTION:
The Vessix System is a highly-differentiated and advanced renal denervation system that features an intuitive push-button interface, a short 30-second treatment time and an over-the-wire, balloon-based approach familiar to most cardiac and vascular specialists. The Vessix System has both CE Mark and TGA approval and is currently available for sale in Europe, the Middle East, Australia, New Zealand and selected markets in Asia. The Vessix System is an investigational device and not available for sale in China. An current analysis of the REDUCE-HTN post market study affirms the device's safety profile and effective treatment for resistant hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Have provided written informed consent
* Are ≥ 18 years and ≤ 75 years of age
* Have a SBP /DBP ≥ 160/90 mm Hg based on an average of three office-based blood pressure readings (seated) measured according to the protocol (≥ 150 mmHg in subjects with Type 2 diabetes)
* On a stable medication regimen with ≥ 3 anti-hypertensive drugs (one of medications should be a diuretic, unless subject has a documented intolerance to diuretics) at maximally tolerated doses and have had no changes to the medication regimen two (2) weeks prior to enrollment
* With a eGFR ≥ 40 ml/min per 1.73m²
* Are willing and able to comply with all study procedures
* With a main renal artery diameter of ≥ 3.5 mm and ≤ 7.0 mm for each of their kidneys
* With a main renal artery without significant stenosis (stenosis defined as < 30%)
* With a renal artery length of ≥ 15 mm

Exclusion Criteria:

* With secondary hypertension
* With Type I Diabetes Mellitus
* Are contraindicated for intravascular contrast material
* Are contraindicated for anticoagulation medications (heparin, aspirin, Angiomax, etc.), analgesic medications (morphine, fentanyl, etc.), anxiolytic medications (alprazolam, lorazepam, diazepam, etc.) or other medications required for an interventional procedure
* With known bleeding or hyper-coagulation disorders
* Have experienced a myocardial infarction, unstable angina pectoris, uncompensated heart failure, or a cerebrovascular accident within six (6) months prior to the screening visit, or have widespread atherosclerosis, with documented intravascular thrombosis or unstable plaques
* Have planned percutaneous vascular or surgical intervention for any reason within the next 6 months
* Have hemodynamically significant valvular heart disease for which reduction of blood pressure would be considered hazardous
* Have an implantable cardioverter defibrillator (ICD) or pacemaker or with a clinically significant abnormal electrocardiogram at time of screening
* Have any serious medical condition, which in the opinion of the investigator, may adversely affect subject safety or the efficacy of the procedure in the study (i.e., subjects with clinically significant peripheral vascular disease, abdominal aortic aneurysm, bleeding disorders)
* Are pregnant, nursing or planning to become pregnant or who are currently taking estrogen or any estrogen-like compound (female participants of childbearing potential must have a negative serum or urine human chorionic gonadotropin (hCG) pregnancy test prior to the procedure)
* Have a known, unresolved history of drug use or alcohol abuse/dependency
* Are currently enrolled in any investigational study wherein subject participation has not been completed
* For any reason, may not be able to understand or comply with instructions
* With only one kidney
* With prior renal denervation procedure
* With prior intervention to right or left renal artery
* With renal artery stenosis as defined by ≥ 30% stenosis confirmed by angiography with two (2) orthogonal views with selective catheterization
* With iliac stenosis requiring intervention at time of procedure and/or within the next six (6) months
* With severe femoral, renal, iliac or aortic calcification that may cause a potential complication at the time of the procedure
* The physician is unable to cannulate the renal artery
* The physician is unable to access the femoral artery by percutaneous means

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The mean reduction of systolic blood pressure measured by office-based blood pressure assessment | at 6-month post procedure

SECONDARY OUTCOMES:
Major adverse event (MAE) rate | at one month post procedure
  Major adverse event (MAE) rate is a composite rate including the following events: All-cause death; Renal failure (eGFR <15 ml/min/1.73m2 or need for renal replacement therapy); Significant embolic event resulting in end-organ damage or intervention to prevent it; Renal artery dissection or perforation requiring intervention;Hospitalization for hypertensive crisis not related to confirmed non-adherence with anti-hypertensive medications; Vascular complications requiring surgical repair, interventional procedure, thrombin injection, or blood transfusion

OTHER OUTCOMES:
Significant new renal artery stenosis rate | 6 months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Yong Huo, MD, Principal Investigator — Beijing University No.1 Affiliated Hospital
Locations (1):
- The Second Affiliated Hosptial of Qingqing Medical Unversity, Chongqing, Chongqing Municipality, China